CLINICAL TRIAL: NCT00630734
Title: Genetic Predictors of Pharmacokinetic Variability in the Drug-drug Interaction Between Darunavir/Ritonavir and Pravastatin: the Role of SLCO1B1 Polymorphisms.
Brief Title: Genetic Predictors of Variability in the Drug-drug Interaction Between Darunavir/Ritonavir and Pravastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0272; TMC114HIV4003
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2012-11-15 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: HIV Infections; Hyperlipidemia
Keywords: HIV; Pravastatin; Darunavir; Ritonavir; Genetic
MeSH Terms: conditions — HIV Infections; Hyperlipidemias | interventions — Pravastatin; Darunavir; Ritonavir; WASH protein, Drosophila

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SLCO1B1 Group 1 (Experimental): Participants with the SLCO1B1 *1A/*1A diplotype; Interventions: pravastatin 40 mg by mouth once daily on days 1-4, washout on days 5-11, darunavir 600 mg and ritonavir 100 mg by mouth twice daily on days 12-18, pravastatin 40 mg by mouth once daily on days 15-18.
  Interventions: Drug: Pravastatin; Drug: Darunavir; Drug: Ritonavir; Other: Washout
- SLCO1B1 Group 2 (Experimental): Participants with the SLCO1B1 *1A/*1B or *1B/*1B diplotype; Interventions: Pravastatin 40 mg by mouth once daily on days 1-4, washout on days 5-11, darunavir 600 mg and ritonavir 100 mg by mouth twice daily on days 12-18, pravastatin 40 mg by mouth once daily on days 15-18.
  Interventions: Drug: Pravastatin; Drug: Darunavir; Drug: Ritonavir; Other: Washout
- SLCO1B1 Group 3 (Experimental): Participants who carry at least one SLCO1B1 *5, *15, or *17 diplotype; Interventions: Pravastatin 40 mg by mouth once daily on days 1-4, washout on days 5-11, darunavir 600 mg and ritonavir 100 mg by mouth twice daily on days 12-18, pravastatin 40 mg by mouth once daily on days 15-18.
  Interventions: Drug: Pravastatin; Drug: Darunavir; Drug: Ritonavir; Other: Washout

INTERVENTIONS:
Drug: Pravastatin — Pravastatin 40 mg by mouth daily on days 1-4
  Other Names: Pravachol
Drug: Darunavir — Darunavir 600mg by mouth twice daily on days 12-18
  Other Names: Prezista
Drug: Ritonavir — Ritonavir 100mg by mouth twice daily on days 12-18
  Other Names: Norvir
Drug: Pravastatin — Pravastatin 40 mg by mouth daily on days 15-18
  Other Names: Pravachol
Other: Washout — Washout (no medication) on days 5-11.

SUMMARY:
Pravastatin (Pravachol) is approved by the Food and Drug Administration (FDA) and is used to treat high cholesterol. Darunavir (Prezista) and ritonavir (Norvir) are approved by the Food and Drug Administration (FDA) to treat HIV infection. When darunavir and ritonavir are given with pravastatin, they can increase the blood levels of pravastatin. The degree of this interaction varies from person to person. The way that darunavir and ritonavir interact with pravastatin may be affected by a person's genetic make-up. Genetic factors (or DNA) are those that people are born with and that make each person unique. Genetic differences are the reason why one person's body traits such as height and hair color are different from another person's body traits. Genetic differences can also affect the way a medication works in the body or the way two medications interact in the body. The purpose of this clinical study is to determine if a person's genetic make-up affects the way darunavir and ritonavir interact with pravastatin in the body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, HIV-negative volunteers

Exclusion Criteria:

* Currently active or chronic cardiovascular, hepatic, renal, pancreatic, gastrointestinal, neurologic, hematologic, psychiatric, metabolic, respiratory, inflammatory, or infectious disease
* Chronic pancreatitis
* History of rhabdomyolysis
* History of statin-associated myopathy
* Active malignancy
* History of significant skin disease, food allergy, drug allergy, dermatitis, eczema, psoriasis
* Pregnancy/breastfeeding
* HIV positive and/or AIDS
* serum creatinine grade 1 or greater (≥ 1.1 x upper limit of laboratory normal range [ULN]);
* hemoglobin grade 1 or greater (≤ 10.9 g/dL);
* platelet count grade 1 or greater (≤ 124.999 x 109/L);
* absolute neutrophil count grade 1 or greater (≤ 1.3 x 109/L);
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) grade 1 or greater (≥ 1.25 x ULN);
* total bilirubin grade 1 or greater (≥ 1.1 x ULN)
* serum lipase grade 1 or greater (≥ 1.1 x ULN)
* serum amylase grade 1 or greater (≥ 1.1 x ULN)
* any other laboratory abnormality of grade 2 or above

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Aquilante, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited from the Denver metro area between March 2008 and September 2009.
Pre-assignment Details: Participants were genetically screened for solute carrier organic anion transporter family, member 1B1 (SLCO1B1) diplotypes as follows: Group 1, *1A/*1A (reference diplotype); Group 2, *1A/*1B or *1B/*1B diplotypes; and Group 3, subjects with at least one copy of the *5, *15, or *17 haplotype.
Groups:
- SLCO1B1 Group 1: SLCO1B1 *1A/*1A diplotype; Pravastatin 40 mg by mouth daily on days 1-4, washout on days 5-11, darunavir/ritonavir 600/100 mg by mouth twice daily on days 12-18, with pravastatin 40 mg added back on days 15-18
- SLCO1B1 Group 2: SLCO1B1 *1A/*1B or *1B/*1B diplotype; Pravastatin 40 mg by mouth daily on days 1-4, washout on days 5-11, darunavir/ritonavir 600/100 mg by mouth twice daily on days 12-18, with pravastatin 40 mg added back on days 15-18.
- SLCO1B1 Group 3: Carriers of at least one SLCO1B1 *5, *15, or *17 haplotype; Pravastatin 40 mg by mouth daily on days 1-4, washout on days 5-11, darunavir/ritonavir 600/100 mg by mouth twice daily on days 12-18, with pravastatin 40 mg added back on days 15-18
Period: Overall Study
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3
Started | 11 | 13 | 8
Completed | 9 | 12 | 7
Not Completed | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3 | Total
Number analyzed (Participants) | 9 | 12 | 7 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 7 | 28
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (11) | 37 (12) | 39 (11) | 36 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 4 | 15
  Male | 7 | 3 | 3 | 13
Region of Enrollment [Number; unit: participants]
  United States | 9 | 12 | 7 | 28

OUTCOME MEASURES:

1. Primary Outcome: Relative Change in Pravastatin Area Under the Plasma Concentration-time Curve (AUC) Over the Dosing Interval
Description: AUC of pravastatin when administered with darunavir/ritonavir divided by AUC of pravastatin when administered alone. The AUC was measured over a 24-hour dosing interval.
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24 hours post-dose
Population: The population analyzed included participants who completed the pravastatin alone phase and the pravastatin + darunavir/ritonavir phase of the study.
Measure: Mean (95% Confidence Interval); unit: ng*hr/ml
Groups:
- SLCO1B1 Group 1: SLCO1B1*1A/*1A diplotype; Pravastatin 40 mg by mouth daily on days 1-4, washout on days 5-11, darunavir/ritonavir 600/100 mg by mouth twice daily on days 12-18, with pravastatin 40 mg added back on days 15-18
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3
Number analyzed (Participants) | 9 | 12 | 7
ng*hr/ml | 1.09 [0.73 to 1.46] | 1.59 [0.83 to 2.36] | 1.75 [0.52 to 2.97]
Statistical Analysis 1: Comparison: SLCO1B1 Group 1 vs SLCO1B1 Group 2 vs SLCO1B1 Group 3; Relative change data were compared between SLCO1B1 diplotype groups using one-way ANOVA (with post-hoc Bonferroni tests); Test type: Superiority or Other; p = 0.43, ANOVA — Threshold of significance was P<0.05

2. Primary Outcome: Relative Change in Pravastatin Maximum Plasma Concentration (Cmax)
Description: Cmax of pravastatin when administered with darunavir/ritonavir divided by the Cmax of pravastatin when administered alone.
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3
Number analyzed (Participants) | 9 | 12 | 7
ng/ml | 1.11 [0.69 to 1.53] | 1.69 [0.83 to 2.55] | 2.32 [0.24 to 4.40]
Statistical Analysis 1: Comparison: SLCO1B1 Group 1 vs SLCO1B1 Group 2 vs SLCO1B1 Group 3; Test type: Superiority or Other; p = 0.28, ANOVA

3. Other Pre Specified Outcome: Darunavir Area Under the Plasma Concentration-time Curve (AUC) Over the Dosing Interval
Description: AUC of darunavir over a 12-hour dosing interval.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3
Number analyzed (Participants) | 9 | 12 | 7
ng*h/ml | 58552 (29442) | 63679 (16985) | 60156 (13909)
Statistical Analysis 1: Comparison: SLCO1B1 Group 1 vs SLCO1B1 Group 2 vs SLCO1B1 Group 3; Test type: Superiority or Other; p = 0.66, ANOVA

4. Other Pre Specified Outcome: Darunavir Maximum Plasma Concentration (Cmax)
Description: Cmax of darunavir over a 12-hour dosing interval
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3
Number analyzed (Participants) | 9 | 12 | 7
ng/ml | 7770 (3483) | 8047 (2023) | 7789 (1467)
Statistical Analysis 1: Comparison: SLCO1B1 Group 1 vs SLCO1B1 Group 2 vs SLCO1B1 Group 3; Test type: Superiority or Other; p = 0.85, ANOVA

5. Other Pre Specified Outcome: Ritonavir Area Under the Plasma Concentration-time Curve (AUC) Over the Dosing Interval
Description: AUC of ritonavir over a 12-hour dosing interval.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3
Number analyzed (Participants) | 9 | 12 | 7
ng*hr/ml | 5239 (3835) | 7178 (3520) | 7907 (3618)
Statistical Analysis 1: Comparison: SLCO1B1 Group 1 vs SLCO1B1 Group 2 vs SLCO1B1 Group 3; Test type: Superiority or Other; p = 0.11, ANOVA

6. Other Pre Specified Outcome: Ritonavir Maximum Plasma Concentration (Cmax)
Description: Cmax of ritonavir over a 12-hour dosing interval
Time Frame: 0,1, 2, 3, 4, 5, 6, 8, 12 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3
Number analyzed (Participants) | 9 | 12 | 7
ng/ml | 844 (708) | 1143 (649) | 1279 (748)
Statistical Analysis 1: Comparison: SLCO1B1 Group 1 vs SLCO1B1 Group 2 vs SLCO1B1 Group 3; Test type: Superiority or Other; p = 0.15, ANOVA

7. Secondary Outcome: Pravastatin Alone: Pravastatin Area Under the Plasma Concentration-time Curve (AUC) Over the Dosing Interval
Description: Dosing interval of 24 hours
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3
Number analyzed (Participants) | 9 | 12 | 7
ng*h/ml | 63 (25.2) | 86.6 (36.3) | 123.4 (80.1)
Statistical Analysis 1: Comparison: SLCO1B1 Group 1 vs SLCO1B1 Group 2 vs SLCO1B1 Group 3; Test type: Superiority or Other; p = 0.22, ANOVA

8. Secondary Outcome: Pravastatin Alone: Pravastatin Maximum Plasma Concentration (Cmax)
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3
Number analyzed (Participants) | 9 | 12 | 7
ng/ml | 27.7 (15.4) | 33.3 (17.1) | 46.2 (38.6)
Statistical Analysis 1: Comparison: SLCO1B1 Group 1 vs SLCO1B1 Group 2 vs SLCO1B1 Group 3; Test type: Superiority or Other; p = 0.67, ANOVA

9. Secondary Outcome: Pravastatin + Darunavir/Ritonavir: Pravastatin Area Under the Plasma Concentration-time Curve (AUC) Over the Dosing Interval
Description: Dosing interval of 24 hours
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3
Number analyzed (Participants) | 9 | 12 | 7
ng*h/ml | 68.4 (37.3) | 106.8 (47.9) | 145.7 (36.9)
Statistical Analysis 1: Comparison: SLCO1B1 Group 1 vs SLCO1B1 Group 2 vs SLCO1B1 Group 3; Test type: Superiority or Other; p = 0.006, ANOVA

10. Secondary Outcome: Pravastatin + Darunavir/Ritonavir: Pravastatin Maximum Plasma Concentration (Cmax)
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SLCO1B1 Group 1 | SLCO1B1 Group 2 | SLCO1B1 Group 3
Number analyzed (Participants) | 9 | 12 | 7
ng/ml | 30.1 (19.7) | 42.4 (23.0) | 52.8 (11.6)
Statistical Analysis 1: Comparison: SLCO1B1 Group 1 vs SLCO1B1 Group 2 vs SLCO1B1 Group 3; Test type: Superiority or Other; p = 0.08, ANOVA

ADVERSE EVENTS:
Groups:
- Pravastatin Alone: Pravastatin 40 mg by mouth daily on days 1-4; Includes 32 participants who received at least one dose of pravastatin 40 mg during days 1-4.
- Darunavir/Ritonavir Alone: Darunavir/Ritonavir 600/100 mg by mouth twice daily on days 12-14; Includes 31 participants who received at least one dose of darunavir/ritonavir during days 12-14.
- Pravastatin + Darunavir/Ritonavir: Darunavir/ritonavir 600/100 mg by mouth twice daily and pravastatin 40 mg by mouth once daily on days 15-18. Includes 28 participants who received at least one dose of darunavir/ritonavir and pravastatin during days 15-18.
Arm/Group | Pravastatin Alone | Darunavir/Ritonavir Alone | Pravastatin + Darunavir/Ritonavir
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 1/28
Other Adverse Events (participants affected / at risk) | 13/32 | 22/31 | 18/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pravastatin Alone (N=32) | Darunavir/Ritonavir Alone (N=31) | Pravastatin + Darunavir/Ritonavir (N=28)
Angioedema (General disorders) | 0 (0) | 0 (0) | 1 (1) — 1 patient experienced grade 2 angioedema (as described by DAIDS criteria). This was not technically SAE, but did require pharmacologic intervention to prevent a more serious reaction.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pravastatin Alone (N=32) | Darunavir/Ritonavir Alone (N=31) | Pravastatin + Darunavir/Ritonavir (N=28)
Headache (General disorders) | 8 (8) | 8 (8) | 6 (6) — Grade 1 per DAIDS criteria.
Fatigue (General disorders) | 2 (2) | 5 (5) | 1 (1) — Grade 1 per DAIDS criteria.
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) — Grade 1 per DAIDS criteria.
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 3 (3) — Grade 1 per DAIDS criteria.
Dizziness (General disorders) | 2 (2) | 0 (0) | 1 (1) — Grade 1 per DAIDS criteria.
Hypoalbuminemia (General disorders) | 3/28 (3) | 3 (3) | 2 (2) — Grade 1 per DAIDS criteria.
Nausea/Vomiting/Dyspepsia/Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 12 (12) | 3 (3) — Grade 1 per DAIDS criteria.
Diarrhea (Gastrointestinal disorders) | 1 (1) | 8 (8) | 13 (13) — Grade 1 per DAIDS criteria.
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) — Grade 1 per DAIDS criteria.
Shoulder/Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) — Grade 1 per DAIDS criteria.

LIMITATIONS AND CAVEATS:
The study included only heterozygous carriers of the SLCO1B1 *15 and *17 haplotypes. Pravastatin urine concentrations were not measured; therefore the impact of darunavir/ritonavir on pravastatin renal clearance was not assessed in this population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication or presentation, the PI will provide the sponsor with at least 60 days for review of a manuscript